CLINICAL TRIAL: NCT06670638
Title: Development of a Novel Endoscopic Index and Patient-reported Outcome Measure for Clinical Trials in Participants With Permanent Ileostomy
Status: Recruiting | Type: Observational
Sponsor: Alimentiv Inc. (Other)
Collaborators: University of Western Ontario, Canada (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); The Cleveland Clinic (Other); OPEN Health (Pharmerit) (Unknown)
Responsible Party: Sponsor
Other Study IDs: HEL01847
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants enrolled in this study will be invited to donate biopsy samples, serum, and/or stool to the Cleveland Clinic Foundation Gastrointestinal Research Biobank. The provision of these samples is optional and not required for this study. The samples and corresponding deidentified data collected for this study will be transferred to the Cleveland Clinic, where they will be processed, stored, and analyzed for future research purposes not related to this study, including investigation of aspects of IBD that may lead to improved treatments and management strategies for individuals affected by IBD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, patients with Crohn's Disease (CD) and permanent ileostomies have been excluded from clinical trials for new treatments. To allow this patient population to be included in clinical trials, outcome and measurement tools are needed. This study aims to develop a Patient Reported Outcome (PRO) and Endoscopic Index (EI) for patients with Crohn's Disease (CD) and permanent ileostomy. The study will enroll about 50 participants and collect videos of endoscopies that are done as part of standard of care. The videos will be centrally read to identify features that represent a broad range of inflammation and will be used to develop the EI. Participants will also be asked to participate in interviews, to understand the symptoms and impacts that are most important to participants for the development of a PRO.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years) with a diagnosis of CD treated surgically with subtotal colectomy/proctocolectomy end ileostomy at least 12 months prior to the scheduled endoscopy procedure.
2. Planning to have an ileoscopy procedure scheduled as part of routine medical care.
3. Be proficient in the English language (ie, ability to read, write, speak, and understand English well enough to take part in the interview process without the aid of an interpreter).
4. Able and willing to participate fully in all aspects of this study.
5. Written informed consent must be obtained and documented.

Exclusion Criteria:

1. End or loop colostomy, end ileostomy for UC, continent ileostomy, ileal pouch anal anastomosis, end ileostomy with mucous fistula, double barrel ileostomy, urostomy, loop ostomy, or any type of end ileostomy not considered permanent at the time of enrolment (with no intent to restore continuity).
2. Peristomal skin complications such as pyoderma gangrenosum, abscess, or any other severe peristomal skin inflammation.
3. Stomal stenosis obviating ileoscopy, known small bowel stricture, major stoma prolapse, symptomatic parastomal hernia, parastomal hernia with subcutaneous loops of small bowel within the hernia, stoma in a crease/poorly fitting applicable resulting in severe peristomal skin irritation, or retracted stoma that prevents endoscopic evaluation.
4. Any actively draining fistula (eg, peristomal or peri-anal).
5. Evidence of a known small bowel stricture on cross-sectional imaging or inability to pass an endoscope within the past 6 months.
6. Known active Clostridoides difficile or other enteric infection.
7. Short bowel syndrome.
8. Predominant symptom(s) arising from a retained rectal stump.
9. Serious underlying disease other than CD that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study procedures or provide nonconfounded descriptions of their CD and ostomy symptom experiences during the interview.
10. Prior enrolment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 participants who meet the inclusion and exclusion criteria will be enrolled in the study. The study population will ideally include approximately equal distributions of participants with disease activity categorized by a central reader as normal, mild, moderate, and severe, according to the VAS assessment. It is not possible to predetermine the number of participants with specific disease activity levels. The distribution of inflammatory disease activity across the study population will be monitored on an ongoing basis and recruitment strategies may be reviewed for opportunities to help maintain a balanced distribution. No more than 10 asymptomatic participants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Develop a PRO instrument for patients with Crohn's Disease and Permanent Ileostomy | through study completion, and average of 1 year
  Concept elicitation interviews focusing on the symptoms and impacts relevant to patients with CD and permanent ileostomy will be conducted and used to develop a PRO. Cognitive interviews will subsequently be conducted to determine respondent comprehension and relevance of the items.
Evaluate the intrarater reliability of 100-mm VAS. | At baseline and 2 weeks
  Central readers will score endoscopy videos using the VAS, on 2 separate occasions at least 2 weeks apart. Intrarater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the intrarater reliability of RAM identified items. | At baseline and 2 weeks
  Central readers will score endoscopy videos for items identified during a RAND/UCLA appropriateness method, on 2 separate occasions at least 2 weeks apart. Intrarater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the intrarater reliability of Rutgeerts score and its component items. | At baseline and 2 weeks
  Central readers will score endoscopy videos using the Rutgeerts Score, on 2 separate occasions at least 2 weeks apart. Intrarater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the intrarater reliability of CDEIS and its component items. | At baseline and 2 weeks
  Central readers will score endoscopy videos using the CDEIS, on 2 separate occasions at least 2 weeks apart. Intrarater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the intrarater reliability of SES-CD and its component items. | At baseline and 2 weeks
  Central readers will score endoscopy videos using the SES-CD, on 2 separate occasions at least 2 weeks apart. Intrarater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the interrater reliability of 100-mm VAS. | At baseline
  Central readers will score endoscopy videos using the VAS, on 2 separate occasions at least 2 weeks apart. Interrater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the interrater reliability of RAM identified items. | At baseline
  Central readers will score endoscopy videos for items identified during a RAND/UCLA appropriateness method, on 2 separate occasions at least 2 weeks apart. Interrater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the interrater reliability of Rutgeerts score and its component items. | At baseline
  Central readers will score endoscopy videos using the Rutgeerts score, on 2 separate occasions at least 2 weeks apart. Interrater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the interrater reliability of CDEIS and its component items. | At baseline
  Central readers will score endoscopy videos using the CDEIS, on 2 separate occasions at least 2 weeks apart. Interrater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Evaluate the interrater reliability of SES-CD and its component items. | At baseline
  Central readers will score endoscopy videos using the SES-CD, on 2 separate occasions at least 2 weeks apart. Interrater reliability will be quantified using ICC, which are equivalent to weighted Kappa statistics in the case of ordinal data.
Develop a novel index using a multiple regression approach with the dependent variables being the VAS and candidate independent variables including items having at least moderate interrater reliability. | through study completion, and average of 1 year
  A prototype index will be created using the VAS for global assessment of severity as the dependent criterion. Prospective validation of the endoscopic index will be performed in a future initiative outside of the scope of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rieder, Principal Investigator — The Cleveland Clinic; Vipul Jairath, Principal Investigator — Western University, Canada
Locations (5):
- United States (3):
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - Washington University in St Louis School of Medicine, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - LHSC - University Campus, London, Ontario